CLINICAL TRIAL: NCT03907774
Title: A Feasibility Study of 12 Weeks of Smartphone-based Health Education Podcasts in Myeloproliferative Neoplasm Patients
Brief Title: MPN Podcast Pilot Study
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00008403
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Myeloproliferative Neoplasm, Unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrolled MPN patients will participate in a podcast intervention via a smartphone app. They will listen to 60 minutes per week of podcasts through this app, which consist of cancer-related health education material. Participants have the option to listen to additional podcasts beyond the 60-minute weekly prescription if they desire. Participation will be tracked through self-report logs. In addition, questionnaires will be administered at baseline, midpoint (week 6), and post-intervention (week 12), which ask about demographics, health information, and satisfaction. The hypothesis is that the smartphone app is feasible for delivering home-based health education podcasts to MPN patients.

DETAILED DESCRIPTION:
Interested patients will complete an eligibility screening using a REDCap link (see eligibility survey). The eligibility screening takes 5-10 minutes to complete.

If ineligible, the participant will be sent an email notification (see study protocol).

If eligible, the potential participant will be sent a link to a video containing a detailed overview of the informed consent as well as a link to sign the informed consent. There will be a place for the participant to type in their electronic signature, which will constitute their consent to participate in the study (see informed consent). After signing the informed consent, participants will be sent an additional email with their study start date, which will fall on the next Monday after signing the informed consent so that all participants begin participating on a Monday. On the day of their study start date, participants will be sent a welcome email as well as a link to complete the baseline self-report measure (listed below) via REDCap.

Within the welcome email, there will be step-by-step instructions for accessing the podcast intervention via a smartphone app. Participants will be asked to view 60 minutes per week of podcasts through a smartphone app. The podcast videos will contain general cancer-related health education material. A total of 60 minutes per week will be prescribed, however, participants will have the ability to view additional videos each week. Furthermore, participants will also track their podcast video viewing each week in a weekly log (see weekly log) by recording each time they view a video, the video that they viewed, and how long they viewed the video.

The investigators will use self-report questionnaires at baseline (week 0), mid-point (week 6), and post-intervention (week 12) administered via REDCap (see baseline, mid-point, and post-intervention surveys). Demographics data and MPN-related health information will be collected at baseline and satisfaction-related data will be collected within the post-intervention questionnaire. Feasibility measures will include acceptability, demand, and practicality.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of essential thrombocythemia, polycythemia vera, or myelofibrosis identified by treating physician
* Have access to a smartphone on a regular basis
* Have access to reliable home internet
* Read and understand English
* 18 years or older

Exclusion Criteria:

* Any planned change in pharmacologic intervention (i.e., new drug, bone marrow transplant) during the study interval (i.e., 12 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group will be compiled of eligible participants recruited through physicians, social media, and other online-based recruitment strategies.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Acceptability of Podcast App: satisfaction survey | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  Acceptability will be measured with a satisfaction survey. Benchmarks for acceptability include greater than or equal to 70% response to the following questions in the survey: 1) satisfaction with the app's content, 2) intending to continue using the app, 3) enjoying using the apps, and 4) recommending it to other MPN patients. The % of participants indicating responses to the four prior questions will be considered "acceptable" if all four questions are responded to with a greater than or equal to 70% response rate.
Demand of Podcast App | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  Demand will be measured using adherence to the podcast prescription. Podcast viewing will be tracked by the smartphone app developers and reported to the Principal Investigator. Adherence benchmarks are defined as an average of greater than or equal to 49 minutes per week of podcast viewing across all participants (i.e., greater than or equal to 70% of prescribed podcasts).
Practicality of Podcast App: participation rate | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  Practicality will be measured through a participation rate greater than or equal to 70%, with completion being defined as completing all three self-report questionnaires.

SECONDARY OUTCOMES:
MPN Total Symptom Burden (severity and symptomology) | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  A 10-item, validated form that calculates total symptom burden score through the MPN Symptom Assessment Form Total Symptom Score. A higher score indicates a worse MPN-specific symptom burden; scores range from 0-100.
Fatigue | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  A single-item fatigue question taken from the MPN Symptom Assessment Form; scores can range from 0-10.
Anxiety | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH Promis) Anxiety Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 36.3-82.7.
Depression | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH Promis) Depression Adult Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 41.0-79.4.
Sleep Disturbance | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH Promis) Sleep Disturbance Adult Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 32.0-73.3.
Sexual Function | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH Promis) Sexual Function consisting of five sub-scales; these scales consist of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; the five sub-scales include vaginal discomfort (score range of 33.2-77.08), lubrication (score range of 30.99-69.26), erectile dysfunction (score range of 30.72-68.47), satisfaction with sex life (score range of 29.59-72.01), and interest in sexual activity (score range of 32.02-76.17).
Pain Intensity: NIH Promis Pain Intensity Adult Short Form | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH Promis) Pain Intensity Adult Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 30.7-71.8.
Global Health | Change from baseline to mid-point (week 6) and post-intervention (week 12)
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH Promis) Global Health consisting of Physical Health and Mental Health sub-scales; these scales consist of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores ranges for physical health are 16.2-67.7, and score ranges for mental health are 21.1-67.6.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huberty J, Eckert R, Puzia M, Laird B, Larkey L, Mesa R. A Novel Educational Control Group Mobile App for Meditation Interventions: Single-Group Feasibility Trial. JMIR Form Res. 2020 Jul 21;4(7):e19364. doi: 10.2196/19364. PMID 32706719